CLINICAL TRIAL: NCT00863434
Title: A Phase II Trial of Clofarabine and Cytarabine to Treat Minimal Residual Disease (MRD) in Acute Myeloid Leukemia
Brief Title: Clofarabine and Cytarabine in Treating Patients With Acute Myeloid Leukemia With Minimal Residual Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Pamela S Becker, Principal Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6858; NCI-2009-01666 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Recurrent Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Congenital Abnormalities; Leukemia, Myeloid, Acute | interventions — Clofarabine; Cytarabine; Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (colony stimulating factor and chemotherapy) (Experimental): Patients receive G-CSF SC QD on days 1-5 and clofarabine IV over 1 hour and cytarabine IV on days 2-5. Beginning approximately 1 month later, patients may receive one additional course of treatment in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: clofarabine; Drug: cytarabine; Biological: filgrastim

INTERVENTIONS:
Drug: clofarabine — Given IV
  Other Names: CAFdA; Clofarex; Clolar
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Biological: filgrastim — Given SC
  Other Names: G-CSF; Neupogen

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as clofarabine and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving clofarabine together with cytarabine may kill more cancer cells.

PURPOSE: This pilot phase II trial is studying how well giving clofarabine together with cytarabine works in treating patients with acute myeloid leukemia with minimal residual disease

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test the ability of clofarabine + ara-C (cytarabine) to eliminate minimal residual (MRD) in acute myeloid leukemia (AML) patients whose bone marrows exhibit complete remission by morphology.

SECONDARY OBJECTIVES:

I. To determine the duration of complete remission after this treatment to minimize MRD.

OUTLINE:

Patients receive filgrastim (G-CSF) subcutaneously (SC) once daily (QD) on days 1-5 and clofarabine intravenously (IV) over 1 hour and cytarabine IV on days 2-5. Beginning approximately 1 month later, patients may receive one additional course of treatment in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years, and then annually for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AML by World Health Organization (WHO) criteria
* Persistence of MRD by flow cytometry (phenotypic blast population detectable at >= 0.1% by flow cytometry despite < 5% blasts by morphology) after initial induction and one to four cycles of cytarabine containing consolidation chemotherapy
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
* Serum creatinine =< 1.0 mg/dL; if serum creatinine > 1.0 mg/dL, then the estimated glomerular filtration rate (GFR) must be > 60 mL/min/1.73m^2 as calculated by the Modification of Diet in Renal Disease equation, as reported by University of Washington Medical Center (UWMC) laboratory system
* Serum bilirubin =< 1.5 x upper limit of normal (ULN)
* Aspartate transaminase (AST)/alanine transaminase (ALT) =< 2.5 x ULN
* Alkaline phosphatase =< 2.5 x ULN
* Capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent
* Female patients of childbearing potential must have a negative serum pregnancy test within 2 weeks prior to enrollment
* Male and female patients must use an effective contraceptive method during the study and for a minimum of 6 months after study treatment

Exclusion Criteria:

* Current concomitant chemotherapy, radiation therapy, or immunotherapy other than as specified in the protocol
* Use of investigational agents within 30 days or any anticancer therapy within 2 weeks before study entry, with exceptions for oral agents such as FMS-like tyrosine kinase 3 (Flt3) Inhibitors or hydroxyurea which will be discontinued prior to the investigational drug regimen; intrathecal treatment within two weeks will also be allowed but not permitted to be given concurrently with investigational regimen
* The patient must have recovered from all acute non-hematological toxicities from any previous therapy
* Have any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney, liver, or other organ system that may place the patient at undue risk to undergo treatment
* Patients with a systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment)
* Pregnant or lactating patients
* Any significant concurrent illness, condition, or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results
* Have had a diagnosis of another malignancy, unless the patient has been disease free for at least 3 years following the completion of curative intent therapy including the following:
* Patients with treated non-melanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia, regardless of the disease-free duration, are eligible for this study if definitive treatment for the condition has been completed
* Patients with organ-confined prostate cancer with no evidence of recurrent or progressive disease based on prostate-specific antigen (PSA) values are also eligible for this study if hormonal therapy has been initiated or a radical prostatectomy has been performed
* Prior allogeneic stem cell transplant
* Prior treatment with clofarabine

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-02; Primary Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Becker, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Colony Stimulating Factor and Chemotherapy)
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Colony Stimulating Factor and Chemotherapy)
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 41.5 [34 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 2
Minimal Residual Disease (blast %) as Assessed by Bone Marrow Flow Cytometry [Median (Full Range); unit: percent of white blood cells] — Percent of white blood cells that are blasts (by flow cytometry).
  percent of white blood cells | 4.35 [4.3 to 4.4]

OUTCOME MEASURES:

1. Primary Outcome: Minimal Residual Disease as Assessed by Bone Marrow Flow Cytometry
Description: Percent of white blood cells that are blasts in the bone marrow post-treatment.
Time Frame: Post-treatment
Measure: Median (Full Range); unit: percent of white blood cells
Arm/Group | Treatment (Colony Stimulating Factor and Chemotherapy)
Number analyzed (Participants) | 2
percent of white blood cells | 1.8 [.2 to 3.4]

2. Primary Outcome: Disease-free Survival
Time Frame: Every 3 months for 2 years, and then annually for 3 years
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Colony Stimulating Factor and Chemotherapy)
Number analyzed (Participants) | 2
months | 6.43 [3.27 to 9.6]

3. Primary Outcome: Overall Survival
Time Frame: Every 3 months for 2 years, and then annually for 3 years
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Colony Stimulating Factor and Chemotherapy)
Number analyzed (Participants) | 2
months | 9.73 [8.27 to 11.2]

ADVERSE EVENTS:
Arm/Group | Treatment (Colony Stimulating Factor and Chemotherapy)
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Colony Stimulating Factor and Chemotherapy) (N=2)
Exacerbation of depression (Psychiatric disorders) | 1 (1)
Left shoulder pain (General disorders) | 1 (1)
Macular Rash (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No